CLINICAL TRIAL: NCT01116128
Title: A Multicenter, Open-label, Phase Ii Study of Dasatinib in Combination With Melphalan and Prednisone (D-MP) in Advanced, Relapsed / Refractory Multiple Myeloma Patients
Brief Title: Dasatinib in Combination With Melphalan and Prednisone to Treat Relapsed and Refractory Multiple Myeloma Patients
Acronym: D-MP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty in enrolling patients
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Prof. Mario Boccadoro, Fondazione Neoplasie Sangue Onlus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-210
Record Dates: First submitted 2010-03-17; First posted 2010-05-04 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Myeloma
Keywords: relapsed/refractory myeloma patients; Progression free survival; Overall survival; dasatinib
MeSH Terms: conditions — Neoplasms, Plasma Cell; Recurrence | interventions — Dasatinib; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- D-MP (Experimental)
  Interventions: Drug: dasatinib; Drug: melphalan; Drug: prednisone

INTERVENTIONS:
Drug: dasatinib — 100 mg QD continuously (from day 1 to day 28)
Drug: melphalan — 0,18 mg/Kg/day from day 1 to day 4 for 6 cycles
Drug: prednisone — 1,5 mg/Kg/day from day 1 to day 4 for 6 cycles

SUMMARY:
Clinically demonstrated efficacy of Melphalan and Prednisone in MM subjects as well as the confirmed inhibitory effect of dasatinib on several tyrosine kinase receptors and pathways implicated in the pathophysiology of MM. Additionally, as a SRC inhibitor, dasatinib plays an important role on bone metabolism through inhibition of osteoclast-mediated bone resorption in vitro. Dasatinib could, thus, be beneficial on bone density of patients on study, through blockage of osteolysis and control of bone lesions.

DETAILED DESCRIPTION:
Primary Objective: To determine whether the combination of dasatinib with melphalan and prednisone provides therapeutic benefits and is safe in patients with relapsed/refractory Multiple Myeloma.

Study design, dose and mode of administration, and duration of treatment: Multicenter, open-label, single arm, two-stage, Phase II study of dasatinib in combination with melphalan and prednisone (D-MP) in advanced, refractory MM patients. The three drugs will be concurrently administered through 6 cycles; each cycle will be 28 days long (1 cycle = 4 weeks), for a total of 24 weeks of treatment. The treatment schedule will be the following:

* Melphalan 0,18 mg/Kg/day from day 1 to day 4 for 6 cycles;
* Prednisone 1,5 mg/Kg/day from day 1 to day 4 for 6 cycles;
* Dasatinib 100 mg QD continuously (from day 1 to day 28). After the 6 cycles of D-MP treatment, Dasatinib will be continuously administered alone as maintenance, until occurrence of progressive disease, unacceptable toxicity or informed consent withdrawal.

This is a two-stage Phase II trial according to Simon with a bivariate endpoint design, by which treatment efficacy and safety are jointly evaluated. This design allows the trial to be early stopped after the first stage if the number of observed partial responses (PR) is inadequate and the number of observed toxicities is too high. In the first stage of the protocol 17 patients are required.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤75 year
2. Karnofsky performance status ≥ 60%
3. Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
4. Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
5. Patient of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped.
6. Patient was previously diagnosed with symptomatic MM based on standard criteria, and has measurable disease, defined as follows:

   * Secretory myeloma: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours;
   * Non-secretory myeloma: > 30% plasma cells in the bone marrow and at least one plasmocytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e., MRI or CT scan).
7. Patient is relapsed or refractory and has received previous regimen containing Thalidomide or Lenalidomide and Bortezomib or even MP (patient is refractory if there is a progression during the last therapy or within 2 months after its completion).
8. Patient has a life-expectancy > 3 months
9. Patient has ≤ Grade 2 peripheral neuropathy within 28 days before enrollment and all acute toxicities from any prior therapy (radiotherapy, chemotherapy or surgical procedures) must have resolved to grade ≤ 2, according to the NCI CTCAE version 3.0 at study entry.
10. Patient has the ability to take oral medication (dasatinib must be swallowed whole)
11. Concomitant Medications:

    - Patient agrees that IV bisphophonates will be withheld for the first 8 weeks of Dasatinib therapy due to risk of hypocalcemia.
12. Patient has the following laboratory values within 28 days before Baseline day 1 of the Cycle 1:

    * Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN)
    * Hepatic enzymes (AST, ALT ) ≤ 2.5 times the institutional ULN
    * Serum Na, K+, Mg2+, Phosphate and Calcium > Lower Limit of Normal (LLN)
    * Calculated or measured creatinine clearance: ≥ 20 mL/minute
    * Hemoglobin, Neutrophil count, Platelets, PT, PTT, Fibrinogen all Grade 0-1
    * Corrected serum calcium ≤ 14 mg/dL ( ≤ 3.5 mmol/L).

Exclusion Criteria:

1. Patients with > 2 previous treatment regimens.
2. Multiple myeloma treatment (ie, chemotherapy, biological, immunotherapy or investigational agent [therapeutic or diagnostic]) administered within 21 days prior to treatment initiation.
3. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
4. Pregnant or breast feeding females.
5. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
6. Use of any other concomitant standard/experimental anti-myeloma drug or therapy
7. Concurrent anticoagulation treatment or medications that directly or durably inhibit platelet function.
8. Malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 5 year. Exceptions: basal cell or non metastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or FIGO Stage 1 carcinoma of the cervix.
9. Concurrent medical condition which may increase the risk of toxicity, including:

   - Pleural or pericardial effusion of any grade
10. Clinically significant cardiac disease (NYHA classification III and IV); any of the following should be considered for exclusion:

    1. Uncontrolled angina, congestive heart failure or MI within (6 months)
    2. Diagnosed congenital long QT syndrome
    3. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
    4. Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
    5. Subjects with hypokalemia or hypomagnesemia, if it cannot be corrected prior to dasatinib administration.
11. History of significant bleeding disorder unrelated to cancer, including:

    1. Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
    2. Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
    3. Ongoing or recent (< 3 months) significant gastrointestinal bleeding.
12. Concomitant Medications, any of the following should be considered for exclusion:

    1. Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to start dasatinib)

       * quinidine, procainamide, disopyramide
       * amiodarone, sotalol, ibutilide, dofetilide
       * erythromycin, clarithromycin
       * chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, zyprasidone
       * cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
    2. The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy. If antacid therapy is needed, the antacid dose should be administered at least 2 hours prior to or 2 hours after the dose of dasatinib.
    3. Patient may not be receiving any prohibited CYP3A4 inhibitors (see Section 8.6 Prohibited therapies-). Refer to Section Prohibited therapies for other concomitant medications you may wish to prohibit based on disease/patient population.
13. Women who:

    1. are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or
    2. have a positive pregnancy test at baseline, or
    3. are pregnant or breastfeeding. Sexually active women of childbearing potential (WOCBP) must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. All WOCBP MUST have a negative pregnancy test prior to first receiving dasatinib. If the pregnancy test is positive, the patient must not receive dasatinib and must not be enrolled in the study.
14. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.
15. Patient that assume anti-arrhythmic drugs or other medicinal products which led to QT prolongation and cumulative high dose anthracycline.
16. Patient has active infectious hepatitis type B or C or HIV.
17. Patient has known intolerance to lactose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Partial response rate is a primary study endpoint. | 4 years
  Evaluation of tumor status will be conducted at screening and anti-tumor treatment efficacy will be assessed at every cycle according to the International Uniform Criteria for Response in MM.
  Safety and tolerability are a co-primary endpoint: incidence of grade 3-4 toxicities will support the decision to move to stage 2, together with PR rate once all the patients accrued to the first stage are evaluable.

SECONDARY OUTCOMES:
Secondary objectives are progression-free survival and overall survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Mario Boccadoro, MD, Principal Investigator — Divisione Universitaria di Ematologia Ospedale Molinette di Torino
Locations (1):
- Mario Boccadoro, Torino, Italy